CLINICAL TRIAL: NCT00175136
Title: A Comparison of the Design of Tibia Stems - Wedge Stem Versus I-beam Stem. A Prospective Randomized Migration- and Bone Density Study on Primary Cemented Knee Implants.
Brief Title: A Comparison of the Design of Tibia Stems in Cemented Total Knee Arthroplasty - Wedge Stem Versus I-beam Stem.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20030239
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2023-01-04 (Actual); Status verified 2010-10

CONDITIONS: Osteoarthritis
Keywords: RSA; DEXA; Gonarthrosis; Knee Arthroplasty; Micromotion of polyethylen liner; Stem arthroplasty design
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I-beam (Active Comparator): I-beam stem design of tibial component for Total Knee Arthroplasty.
  Interventions: Device: Maxim TKA
- wedge (Active Comparator): Wedge stem design of tibial component for Total Knee Arthroplasty.
  Interventions: Device: Maxim TKA

INTERVENTIONS:
Device: Maxim TKA — Operation with Total Knee Arthroplasty and either an I-beam stem or a wedge stem of the tibial component.
  Other Names: Biomet Merck: Maxim TKA

SUMMARY:
The purpose of this study is to compare the early migration and periprosthetic bone changes of two cemented total knee arthroplasties with different tibial stem design. Only the tibial prostheses plateau varies in that one is an wedge-shaped stem and the other is a I-shaped stem.

DETAILED DESCRIPTION:
Around 4% of total knee arthroplasties (TKA) are revised 15 years after the primary operation, most due to loosening of the implant. About 70 % TKA are fixed with bone cement and in general the results after total knee arthroplasty are excellent and with the existing technique about 95% well functioning prostheses can be expected 10 years post surgery. The most serious late complication to surgery is aseptic loosening of the implants; and this remains one of the main courses of failure of both uncemented and cemented total knee implants.

Implant design, method of fixation and the bone mass density has a large influence on implant stability. Fixation of the tibia base plates in total knee arthroplasty can be obtained by different designs of anchorage in the tibia e.g. central round stems, fins and pegs. The smaller the tibia stem; the lesser amount of bone is lost at implantation and following revisions rendering probable a time gain before secondary arthrodesis is necessary. The tibia stem cannot be to tiny either because it has to be able to resist the load of shearing forces naturally presented by the knee kinetics.

In this project we are using modularly tibia components with a central wedge- and I-beam shaped stem respectively. Both type of prosthesis are consolidated in the bone by bone cement applied under the base-plate while the stem is fixed press-fit (without cement) in the proximal tibia.

The purpose of this study is to compare the early migration of two cemented total knee implants with different tibial stem design by RSA (radio stereophotogrammetric analysis). Furthermore, we will make research into the periprosthetic bone and it's changes after surgery using DEXA. Finally the extend of the expected micromovements between the polyethylene liner and the metal backing of the titanium plateau will be compared and taken into account with the results.

Tibia wedge stems are exposed to the greatest load test by shearing forces while block stems are bearing the greater load with compression and some scientists therefore speculate that block-designs are better than wedge-designs. This project is set up to explain the theoretical speculations about design and implant survival. The durability of the implants have been tested in account of fatigue and durability in a 80-20 test and they're both able to resist 4-6 times bodyweight. Furthermore, the polyethylene is produced by direct compression molding making it very resistant to wear.

To evaluate both the implant-bone micromotions and the polyethylene-implant micromovements metal markers have been placed on the implant prior to surgery and furthermore into the tibial bone and into the tibial polyethylene intra-operatively allowing us to evaluate stereo x-rays by a photogrammetric computer analyses called RSA at the Orthopaedic Center, Aarhus University Hospital. Follow-up stereo x-rays will be scheduled for 1 week, 3 months, 6 month, 1 years and 2 years post-surgery. Periprostetic bone density will be evaluated at 1 week, 1 year and 2 years upon inclusion at the Orthopaedic Center, Aarhus University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one- or double-sided primary knee arthrosis.
* Patients with a sufficient bone quality for implantation of knee prosthesis.
* Informed and written patient consent.

Exclusion Criteria:

* Patients with neuromuscular or vascular diseases in the affected leg.
* Patients who peroperatively are estimated unsuitable for knee arthroplasty e.g. due to bone cysts or dilution of the bone mass.
* Patients who use non-steroid anti-inflammatory drugs (NSAID) and cannot refrain from taking them postoperatively (this includes COX-2-inhibitors).
* Patients with osteoporosis estimated from the preoperative x-ray or former diagnosis of osteoporosis.
* Patients with knee arthrosis following fracture sequelae.
* Women, who are pregnant or are at risk of getting pregnant throughout the 2 year follow-up.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2005-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Tibial component migration evaluated by RSA. | post-operative, three months, six months, one year, two years
Periprosthetic bone changes evaluated by DEXA. | post-operative, one year, two years

SECONDARY OUTCOMES:
Micromotion of the modular polyethylene liner in both type prostheses evaluated by RSA. | post-operative, three months, six months, one year, two years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD, Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Tage-Hansens Gade 2, 8000 Aarhus C, Denmark.
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark